CLINICAL TRIAL: NCT02271503
Title: A Study to Assess the Pharmacokinetics and Pharmacodynamics of a Single Dose of IPX203 in Patients With Advanced Parkinson's Disease
Brief Title: A Study to Assess the PK and Pharmacodynamics of IPX203 in Patients With Advanced Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPX203-B14-02
Record Dates: First submitted 2014-10-13; First posted 2014-10-22 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Other): Subject received a single dose of IPX203 180 mg and/or IPX203 270mg in Period 1, a single dose of CD-LD IR in Period 2, and a single dose of Rytary 145 mg and/or Rytary 195 mg in Period 3.
  Interventions: Drug: CD-LD IR; Drug: IPX203 180 mg; Drug: IPX203 270 mg; Drug: Rytary 195 mg; Drug: Rytary 145 mg
- Sequence 2 (Other): Subject received a single dose of a single dose of CD-LD IR in Period 1, a single dose of Rytary 145 mg and/or Rytary 195 mg in Period 2, and a single dose of IPX203 180 mg and/or IPX203 270mg in Period 3.
  Interventions: Drug: CD-LD IR; Drug: IPX203 180 mg; Drug: IPX203 270 mg; Drug: Rytary 195 mg; Drug: Rytary 145 mg
- Sequence 3 (Other): Subject received a single dose of a single dose of Rytary 145 mg and/or Rytary 195 mg in Period 1, a single dose of IPX203 180 mg and/or IPX203 270mg in Period 2, and a single dose of CD-LD IR in Period 3.
  Interventions: Drug: CD-LD IR; Drug: IPX203 180 mg; Drug: IPX203 270 mg; Drug: Rytary 195 mg; Drug: Rytary 145 mg

INTERVENTIONS:
Drug: CD-LD IR — CD-LD IR containing 25 mg carbidopa and 100 mg levodopa
  Other Names: Sinemet
Drug: IPX203 180 mg — IPX203 containing 45 mg carbidopa and180 mg levodopa
  Other Names: CD-LD ER 180 mg
Drug: IPX203 270 mg — IPX203 containing 67.5 mg carbidopa and 270 mg levodopa
  Other Names: CD-LD ER 270 mg
Drug: Rytary 195 mg — Rytary 48.75Mg-195Mg Extended-Release Capsule
Drug: Rytary 145 mg — Rytary 36.25Mg-145Mg Extended-Release Capsule

SUMMARY:
This is a randomized, open-label, rater-blinded, multicenter, 3-treatment, 3 period, single-dose crossover study. Approximately 51 qualified immediate-release (IR) CD-LD-experienced advanced Parkinson's disease patients will be randomized to 1 of 3 dosing sequences.

Objectives:

* Assess the pharmacodynamics and pharmacokinetics (PK) of IPX203 (carbidopa and levodopa) in subjects with advanced Parkinson's disease.
* Characterize the safety of IPX203 in subjects with advanced Parkinson's disease.

DETAILED DESCRIPTION:
IPX203 contains two different drugs called levodopa and carbidopa in one capsule.

* levodopa turns into a material called 'dopamine' in your brain. The dopamine helps to improve the symptoms of your Parkinson's disease.
* carbidopa belongs to a group of medicines called 'aromatic amino acid decarboxylase inhibitors'. It helps levodopa work more effectively by slowing the speed at which levodopa is broken down in your body.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects diagnosed with idiopathic PD with motor complications, who are currently being treated chronically with stable regimens of CD-LD.

Requiring at least 400 mg but not more than 1600 mg LD per day during the waking hours; and at least 100 mg but not more than 250 mg LD from IR CD-LD for the first morning dose.

Dosing frequency of IR CD-LD of at least 4 times daily excluding nighttime dosing.

Have an average of at least 2 hours per day "off" time during the waking hours and at least 1 hour "off" time per day, based on the PD diary collected for 3 consecutive days prior to Visit 1.

Exclusion criteria:

Have used first morning dose of controlled-release (CR) CD-LD or Rytary for at least 4 weeks prior to Visit 1.

Female subjects who are currently breastfeeding or lactating.

Had prior functional neurosurgical treatment for PD (ablation or deep brain stimulation) or if such procedure(s) are planned or anticipated during the study period.

Allergic to study drugs

History of medical conditions or of a prior surgical procedure that would interfere with LD absorption, such as gastrectomy or small-bowel resection.

History of peptic ulcer disease or upper gastrointestinal hemorrhage.

History of narrow angle glaucoma.

History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias; neuroleptic malignant syndrome; or nontraumatic rhabdomyolysis.

History of psychosis.

Employees or family members of the Investigator, study site, or Sponsor.

Subjects who, in the opinion of the clinical investigator, should not participate in the study.

Based on clinical assessment, subject does not adequately comprehend the terminology needed to complete the PD diary.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
"Off" time per the Assessment of Subject's Motor State | Up to 10 hours

SECONDARY OUTCOMES:
Duration of effect estimated using the timepoint at which an improvement of at least 4 points in the MDS-UPDRS Part III score from predose is first observed and continuing until the timepoint at which the improvement is no longer observed | Up to 10 hours
Change from predose value in the number of finger-taps at each timepoint | Up to 10 hours

OTHER OUTCOMES:
Number of Participants with Adverse Events | Screening through end of study approximately 6 weeks per subject
Maximum concentration (Cmax) | Up to 10 hours
Area under the curve (AUC) | Up to 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (11):
- United States (11):
  - Muhammad Ali Movement Disorder Center (MAMDC), Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - University of South Florida Parkinson's Disease and Movement Disorder Center, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - QUEST Research Institute, Farmington Hills, Michigan
  - Duke University Movement Disorders Clinic, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No